CLINICAL TRIAL: NCT05074706
Title: Evaluation of the Immune Response to Sars-Covid-19 (Cov-2) Vaccines in Haematological Patients: Prospective Single Center Study
Brief Title: Evaluation of the Immune Response to Sars-Covid-19 Vaccines in Haematological Patients: Prospective Single Center Study
Acronym: Hema-C19-Vax
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: San Gerardo Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Hema-C19-Vax
Record Dates: First submitted 2021-10-05; First posted 2021-10-12 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Hematologic Diseases
Keywords: serocoversion; COVID vaccination; cellular immunity; Sars-Cov-2 IgG antibodies; QuantiFERON-SARS-CoV-2 test
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: IgG antibodies to Sars-Cov-2 — Samples will be collected between 30 and 60 days after second vaccine dose.
  Other Names: Blood serum SARS-CoV-2 IgG
Biological: QuantiFERON SARS-CoV-2 test — Samples will be collected within 9 months after completion of the vaccination series
  Other Names: Plasma INF-γ

SUMMARY:
The main objective of this study is to investigate the humoral immune response to COVID-19 vaccines in haematological patients, by testing SARS-CoV-2 seroconversion

DETAILED DESCRIPTION:
This single-center prospective study will enroll approximately 700 hematologic patients who access to Haematological Division (San Gerardo Hospital, Monza, Italy) in order to perform their routine blood tests to monitor their hematological conditions. Evaluation of Sars-Cov-2 IgG specific antibodies will be performed on left-over biological material (serum or plasma) collected during routine blood tests run between 30 and 60 days after the administration of the second vaccine dose.

Furthermore, in each patient who has failed seroconversion (absence of specific antibodies for circulation), his cellular immune response will be assessed using an additional blood sample collected during routine blood tests.

These samples will be collected within 9 months of the completion of the vaccination series and will be used to evaluate the plasma INF-γ release using QuantiFERON SARS-CoV-2 test.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated EC-approved informed consent
* Hematological disease defined according to World Health Organization (WHO) criteria
* Female or male, 18 years of age or older
* ECOG performance status 0-3
* Willingness and ability to comply with routine clinical practice and study procedures
* Regular vaccination against SARS-CoV-2 according to Italian Haematological Society (SIE) guidelines/recommendations (Version 2.0, 20 April, 2021).
* Routine blood test planned between 30 and 60 days after administration of the second vaccine dose according to regular hematological follow up.
* Routine blood test planned no later than 9 months after the completion of the vaccination series (only in case of absence of circulation specific antibodies).

Exclusion Criteria:

* Preventive vaccination against SARS-CoV-2 not administered according to Italian Haematological Society (SIE) guidelines/recommendations (Version 2.0, 20 April, 2021)
* Evidence of previous infection with the SARS-Cov-2 virus.
* Routine blood test not planned between 30 and 60 days after administration of the second vaccine dose.
* Routine blood test not planned within 9 months after the completion of the vaccination series (only in case of absence of circulation specific antibodies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Haematological patients followed at the Haematological Division, San Gerardo Hospital, Monza, Italy
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Rate of seroconversion in hematological patients who received a mRNA SARS-CoV-2 vaccine | Between 30 and 60 days after the administration of the second vaccine dose
  Seroconversion is defined as a post-vaccination SARS-CoV-2 IgG antibody titer >33.8 Binding Anticorpal Unit (BAU)/ml.

SECONDARY OUTCOMES:
To compare the seroconversion rate in haematological patients versus healthy subjects. | Between 30 and 60 days after the administration of the second vaccine dose
  Time adjusted rate of seroconversion after vaccination in hematological patient and healthy population.
To correlate the rate of seroconversion in hematological patients to the specific haematological diseases. | Between 30 and 60 days after the administration of the second vaccine dose
  Rate of seroconversion per type of haematological condition
To correlate the rate of seroconversion to previous therapies | Between 30 and 60 days after the administration of the second vaccine dose
  Rate of seroconversion per specific treatment.
To assess the efficacy of vaccine by estimating how many patients will be infected by SARS-CoV-2 in the 9 months after the administration of the second vaccine dose. | Within 9 months after the administration of the second vaccine dose
  Rate of patients with a positive RT-PCR-SARS-CoV-2 test in the 9 months after the administration of the second vaccine dose
To analize T-cell response in those patients who will result negative for specific antibodies anti-Sars-Cov-2 after two doses of mRNA SARS-Cov-2 vaccination | Within 9 months after the administration of the second vaccine dose
  Rate of patients with a positive QuantiFERON-SARS-CoV-2 test after the demonstration of seroconversion failure until the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gambacorti Passerini, Professor, Study Director — San Gerardo Hospital
Locations (1):
- San Gerardo Hospital, Monza, Lombardy, Italy